CLINICAL TRIAL: NCT02369861
Title: A Randomized, Masked, Active Placebo-controlled Phase 1 Study of Amnion-derived Cellular Cytokine Solution (ACCS) Eye Drops in the Treatment of Dry Eye
Brief Title: Study of ST266 Eye Drops in Treating Dry Eye
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Noveome Biotherapeutics, formerly Stemnion (Industry)
Collaborators: U.S. Navy Bureau of Medicine (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ST-05-14
Record Dates: First submitted 2015-01-14; First posted 2015-02-24 (Estimated); Last update posted 2019-05-13 (Actual); Status verified 2019-05

CONDITIONS: Dry Eye Syndrome
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ST266 (Experimental): Eye drops
  Interventions: Drug: ST266
- Artificial tears (Placebo Comparator): Refresh lubricant eye drops
  Interventions: Drug: Refresh Lubricant Eye Drops

INTERVENTIONS:
Drug: ST266 — Topical ocular application 4 times per day
  Arms: ST266
Drug: Refresh Lubricant Eye Drops — Topical ocular application 4 timer per day
  Arms: Artificial tears

SUMMARY:
Subjects with moderate-to-severe Dry Eye by symptoms will be screened including history, ophthalmic examination to include the status of their ocular structure and function and evaluation of tear production. Blood will be blood drawn for complete blood count and chemistry panel. They will also have a urinalysis and pregnancy test in women of child-bearing potential.

Subjects will have a two week "run-in" period in which they use artificial tears. If their Dry Eye signs and symptoms do not improve significantly, they will be enrolled and will receive study drug.

Safety evaluation includes assessment of the structure and function of the eyes including retina examination and corrected visual acuity.

Subjects who meet the inclusion and exclusion criteria will be randomly assigned to one of two treatment arms, ST266 or "artificial tears" eye drops. The randomization scheme is 1:1 ST266:artificial tears. Subjects will self-administer their eye drops four times each day.

Subjects will be seen in the office of the ophthalmologist/optometrist at baseline (week zero), one week, three weeks, six weeks and ten weeks. Eye examination will be done at each visit. The baseline eye tests and lab work will be repeated after the treatment phase of the study at the end of week six. Following 6 weeks of treatment, the subjects will be followed for 4 additional weeks.

DETAILED DESCRIPTION:
Subjects with moderate-to-severe Dry Eye judged by symptoms will be screened following signing of informed consent. Screening will involve history and physical examination including ophthalmic examination with dilated fundus exam to assess the status of their ocular structure and function, and evaluation of tear production and damage caused by clinically significant Dry Eye. Blood will be blood drawn for complete blood count, chemistry panel including serum glucose, blood urea nitrogen, electrolytes, creatinine, liver function studies including total and direct bilirubin, alkaline phosphatase, alanine transaminase (ALT), aspartate transaminase (AST), albumin, and total protein. They will also have a urinalysis. Pregnancy test will be performed in women of child-bearing potential.

Subjects will have a two week "run-in" period in which they use artificial tears. Those subjects in whom corneal staining is 2 or more (on a scale of 0-4), Dry Eye symptom score on the OSDI is 25-75 after two weeks of using artificial tears four times per day, and laboratory test results within the accepted ranges will be enrolled and will receive study drug, Those subjects in whom dry eye symptoms improve sufficiently (OSDI drops below 25) and/or corneal staining is reduced from 2 or more to less than 2, or have laboratory test results outside the accepted ranges will not be enrolled.

Safety evaluation includes assessment of the structure and function of the eyes including conjunctival and corneal tissues. Corrected visual acuity will be measured at every visit. Patient comfort will be assessed after administration of the study drug and at every visit. A retina examination will be performed before and after the treatment period. Slit lamp exam including the cornea, conjunctiva, anterior chamber, iris, eye lids and lashes will be performed at every visit. Special testing will include fluorescein staining of the cornea, lissamine green staining of the conjunctiva, endothelial cell analysis, Schirmer tear production, and intraocular pressure measured on all subjects.

Subjects who meet the inclusion and exclusion criteria will be randomly assigned to one of two treatment arms, ST266 or "artificial tears" eye drops. ST266 and artificial tears eye drops will be supplied by Stemnion, and both personnel and subjects will be trained in its use. The treatment will be prepared in a coded container such that the subject and physician are masked as to the treatment. One treatment arm will receive ST266 eye drops in both eyes and the other treatment arm will receive artificial tears eye drops in both eyes. Treatment arms will be assigned by random. The randomization scheme is 1:1 ST266:artificial tears. Subjects will self-administer their eye drops four times each day. Subjects will be asked to keep a study diary of when they place the study medication in their eyes.

Subjects will be seen in the office of the ophthalmologist/optometrist at baseline (week zero), one week, three weeks, six weeks and ten weeks. Eye examination will be done at each visit. Each subject will complete a patient questionnaire on their symptoms of Dry Eye. The baseline eye tests and lab work will be repeated after the treatment phase of the study at the end of week six. Following 6 weeks of treatment, the subjects will be followed for 4 additional weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects ages 18 years and older.
2. Subjects with symptoms and signs of Dry Eye for > four months supported by previous clinical diagnosis or self-reported history.
3. Visual acuity corrected 20/40 or better in each eye.
4. If wearing contact lenses, subjects must be willing to refrain from wearing the contact lenses during the study (including washout period).
5. Score of 25-75 on the Ocular Surface Disorder Index (OSDI) questionnaire.
6. Corneal staining of grade 2 or more anywhere on the cornea (scale 0-4).

Exclusion Criteria:

1. Pregnant or breast feeding.
2. Anterior segment disease other than Dry Eye which in the opinion of the investigator would confound the study.
3. Macular and neovascular eye diseases
4. History of corneal surgery or LASIK (laser in situ keratomileusis) surgery in either eye within the past year.
5. Use of cyclosporine, steroid eye drops, serum eye drops, or any other eye medication (except for artificial tears) or experimental drug within the past 30 days.
6. Subjects with glaucoma or in whom glaucoma is suspected.
7. Use of anticholinergic drugs, antihistamines, beta-blockers, or tricyclic anti-depressants within the past 30 days.
8. Asymmetric punctal plugs or punctal cauterization within the past three months.
9. History of Stevens-Johnson disease, ocular cicatricial pemphigoid, alkali burn of the eye, or graft-versus-host disease.
10. Immune compromise for any reason.
11. Kidney or liver function studies >2x the upper limit of normal.
12. Symptomatic abnormalities od the lid.
13. History of cancer within the past 5 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-03; Primary Completion 2015-10 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Corneal staining with fluorescein | Change in degree of staining at 6 weeks
  National Eye Institute Scoring System: 0=none, 1=mild, 2=moderate, 3=severe

SECONDARY OUTCOMES:
Lissamine staining | Change in degree of staining from baseline at 6 weeks
  Lissamine green staining of the conjunctiva
Endothelial cell count | Change from baseline at 6 weeks
  Endothelial cell counts
Intraocular pressure | Change in pressure from baseline at 6 weeks
  Pressure measured by tonometry
Tear volume | Change in tear volume from baseline at 6 weeks
  Schirmer tear production test
Assessment of structure and function of the eye | Change from baseline at 6 weeks
  Change in corrected visual acuity
Assessment of Ocular Surface Disease Index (OSDI) | 6 weeks
  Subject will compete OSDI questionnaire at baseline and at 6 weeks

OTHER OUTCOMES:
Tear osmolarity | Change from baseline at 6 weeks
  Tear osmolarity (osmoles/liter) measured at baseline and after 6 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Steed, MD, Study Director — Noveome Biotherapeutics, formerly Stemnion; Kathy Kelley, OD, Principal Investigator — Price Vision Group
Locations (1):
- Price Vision Group, Indianapolis, Indiana, United States